CLINICAL TRIAL: NCT06321887
Title: A Pilot Study to Assess the Efficacy and Tolerability of Reduced Dose Oral Iron in the Treatment of Iron Deficiency Anaemia in Inflammatory Bowel Disease Patients.
Brief Title: EffiCacy and sAfEty of Low doSe orAl iRon for Anaemia in IBD
Acronym: CAESAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5155
Record Dates: First submitted 2024-02-14; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Disease; Iron Deficiency Anemia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: This is an adaptive, open label study to compare the efficacy and tolerability of 8 weeks of low dose oral iron, in the treatment of iron deficiency anaemia in patients with inflammatory bowel disease (IBD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAGE 1 (Experimental): The first stage shall recruit 10 patients and is used to assess the incidence of oral iron related toxicity.
  Patients will be prescribed:
  • Ferrous fumarate syrup 2.5ml/70mg (22.5mg elemental iron) daily for 8 weeks.
  If patients experience toxicity (defined as symptoms not tolerated by the patient), the trial medication would be stopped and IV Iron treatment given.
  If toxicity occurs in 2 or more patients where we have to stop treatment, we will continue to recruit 30 patients only to the Ferrous fumarate syrup 2.5ml/70mg (22.5mg elemental iron) daily for 8 weeks. If the toxicity is acceptable and the Hb improves, we will continue to recruit to 22.5mg oral iron/day.
  If the toxicity is acceptable but there is no improvement in haemoglobin the next patients will be recruited to stage 2.
  Interventions: Drug: Ferrous fumarate syrup 2.5ml/70mg (22.5mg elemental iron)
- STAGE 2 (Experimental): Ten subjects each will then be sequentially assigned to one of the following groups:
  * Ferrous fumarate syrup 5ml/140mg (45mg elemental iron) daily for 8 weeks.
  * Ferrous fumarate syrup 5ml/140mg twice daily (90mg elemental iron) for 8 weeks.
  If 2 or more patients experience toxicity at Ferrous fumarate syrup 5ml/140mg (45mg elemental iron) or Ferrous fumarate syrup 5ml/140mg twice daily (90mg elemental iron) we will reduce the dose to the previous level of Ferrous fumarate syrup 2.5ml/70mg (22.5mg elemental iron) and continue to recruit.
  30 patients shall be used to estimate the change in haemoglobin between baseline and the final analysis point.
  If no dose reduction is required, only the last 20 patients shall be used to assess haemoglobin.
  The overall endpoint is the haemoglobin level.
  Interventions: Drug: Ferrous fumarate syrup 2.5ml/70mg(45mg elemental iron); Drug: Ferrous fumarate syrup 2.5ml/70mg (90mg elemental iron)

INTERVENTIONS:
Drug: Ferrous fumarate syrup 2.5ml/70mg (22.5mg elemental iron) — Ferrous fumarate syrup 2.5ml/70mg (22.5mg elemental iron) daily for 8 weeks (N=10).
  Arms: STAGE 1
Drug: Ferrous fumarate syrup 2.5ml/70mg(45mg elemental iron) — Ferrous fumarate syrup 5ml/140mg (45mg elemental iron) daily for 8 weeks (N=10).
  Arms: STAGE 2
Drug: Ferrous fumarate syrup 2.5ml/70mg (90mg elemental iron) — Ferrous fumarate syrup 5ml/140mg twice daily (90mg elemental iron) for 8 weeks (N=10).
  Arms: STAGE 2

SUMMARY:
Iron deficiency anaemia (IDA) is common in inflammatory bowel disease (IBD). However, although iron is commonly prescribed, the amount of elemental iron needed to achieve clinical efficacy, and the optimal method of supplementation, are under debate. This pilot study aims to investigate the efficacy and safety of low dose and standard dose oral iron preparations for the treatment of IDA in patients with IBD.

DETAILED DESCRIPTION:
BACKGROUND:

Anaemia, particularly iron-deficiency anaemia, is a common complication of inflammatory bowel disease (IBD). The prevalence of anaemia (6-74%) and iron deficiency (36-90%) varies widely among reported studies. The predominant cause of iron deficiency in IBD is intestinal blood loss but other factors such as malabsorption and reduced intake may also play a role. Thus, the need for iron supplementation is an often encountered clinical problem in IBD. Although iron is commonly prescribed, the amount of elemental iron needed to achieve clinical efficacy, and the optimal method of supplementation, are under debate. As intravenous (IV) iron supplementation has become safer, calls for increased utilization have appeared. However, there are significant cost implications to using IV iron. On average, a 1-month supply of oral ferrous sulfate costs $12, in comparison with approximately $600-$700 for a treatment cycle of (IV) iron sucrose, excluding the cost of IV administration.

Overall, the comparative studies of IV vs. oral iron do not demonstrate a significant difference in haemoglobin repletion favouring IV iron therapy. Haemoglobin concentrations were similar at the end of treatment in all studies. A single study suggested a superiority for IV iron with a haemoglobin increase greater than 2 g/dl in 47% of the patients on oral iron compared with 66% on IV iron (P = 0.07). However, this could be accounted for by a high withdrawal rate (24%) in the oral iron group. In the largest comparative study, of 196 subjects, median haemoglobin improved similarly, from 8.7 to 12.3 g/dl in the IV group and from 9.1 to 12.1 g/dl in the ferrous sulfate group (P = 0.70). Thus, intravenous iron appears no more effective than oral iron in repletion of iron status as the rate-limiting step appears to be synthesis of red cells, which is not accelerated by IV iron delivery.

The main reason behind the preference of IV iron over oral iron is based on the concern that oral iron may exacerbate IBD. An often-cited study investigating whether oral iron worsens IBD in comparison with IV iron assessed disease activity in 19 IBD patients, 11 with CD and 8 with UC, randomized to either oral ferrous fumarate or IV iron sucrose over a 14-day period. Although the authors argued that disease activity was worsened by oral iron therapy, their use of numerous unconventional assessments weakens this conclusion. The trial was done as a crossover study with a minimum 6-week washout period, so the previous drug therapy may have affected the results. The number of subjects with IBD was small (N = 19). The authors created a synthesized overall disease activity score by combining UC and CD scales and also reported on subscales within activity indexes to identify significant differences. When the two groups were compared, however, there was no statistically significant difference in the overall synthesized disease activity score.

Another factor associated with intolerance of oral iron may be related to the dose of elemental iron administered. In order to maintain iron balance, adult men need to absorb 1-1.5 mg/d, menstruating women need 1-3 mg/d, and pregnant women need approximately 4-5 mg/d. Based on this, the recommended daily allowance of elemental iron is about 8 mg in adult men and postmenopausal women, 18 mg in premenopausal women, and 27 mg in pregnant women. However, most studies investigating the efficacy of oral iron have used a typical dose of 150-200mg/d of elemental iron, 10-20 fold in excess of the recommended daily allowance. Because of the 20% incidence level of intolerance at these conventional doses of elemental iron, recent studies have investigated the efficacy and side effects associated with low-dose oral iron supplementation. A study in the elderly (age >80) randomised 90 patients with iron-deficiency anaemia to 15, 50, or 150 mg of daily oral elemental iron over 2 months. All three dosage groups experienced a similar, statistically significant increase in haemoglobin after 2 months. These studies have not been done in IBD.

This pilot study aims to investigate the efficacy and safety of low dose and standard dose oral iron preparations.

HYPOTHESIS:

Low dose oral iron is effective and safe in the treatment of iron deficiency anaemia in inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to participate in the study and has signed the informed consent.
* Patients aged 18-80 years.
* Patients diagnosed with Crohn's disease or ulcerative colitis diagnosed by conventional clinical, radiological and histological criteria.
* Remission or active disease.
* Haemoglobin level 7-13 g/dL men, 7-12 g/dL women and ferritin <30, normal B12 and folate (or ferritin <100 but iron sats <16 in the presence of inflammation defined as CRP>5mg/L, faecal calprotectin>250 microgram/g and presence of endoscopic inflammation).

Exclusion Criteria:

* Patients under 18 or unable to give informed consent.
* Patients with advanced liver disease.
* Patients with advanced renal disease with eGFR<45ml/min
* Previous intolerance to even low doses of oral iron
* Patients with severe cardiovascular disease defined as previous unstable angina and or previous MI without intervention.
* Participation in other trials in the last 3 months.
* Serious inter-current infection or other clinically important active disease (including renal and hepatic disease) and recently diagnosed gastrointestinal tract cancers
* Pregnant, post-partum (<3months) or breast feeding females
* Erythropoietin therapy.
* Recent blood transfusion within 30 days.
* Recent iron infusion within 30 days.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in haemoglobin concentration from baseline to week 8. | 8 weeks
  Measured using serum haemoglobin concentration measured in g/L, taken at week 0 and week 8.

SECONDARY OUTCOMES:
Assessment of iron stores at baseline and week 8 | 8 weeks
  Measured using serum ferritin values measured in ug/L taken at week 0 and week 8.
Assessment of faecal calprotectin at baseline and week 8 | 8 weeks
  Measures on a continuous numeric scale ranging from 21ug/g to 2099ugug. Values outside these thresholds reported as <20ug/g to >2100ug/g.
Assessment of IBD severity. For ulcerative colitis this will be done using simple colitis clinical activity index (SCCAI). Values calculated at week 0 and week 8. | 8 weeks
  SCCAI measured from 0-19 on a continuous numeric scale.
Assessment of IBD severity. For Crohn's disease (or IBD-unclassified) the Harvey Bradshaw Index (HBI) will be used. Values calculated at week 0 and week 8. | 8 weeks
  HBI measured from 0-28 on a continuous numeric scale.
Assessment of quality of life using the IBD-QUK score at baseline and week 8 | 8 weeks
  IBD-QUK measured from 0-96 on a continuous numeric scale, then expressed as a percentage from 0-100%.
Assessment of patient global assessment of symptom severity by visual analogue score at baseline and week 8. | 8 weeks
  A series of eight questions, each comprising a score. The higher the sum of scores, the more severe the symptom profile. Question one pertains to bowel frequency (total number of stools per week), questions two through eight refer to specific gastrointestinal complaints, the severity of which are scored by placing a marker on a 10cm visual scale - the total length of the line marked denotes the severity score for each question.
Assessment of fatigue at baseline and week 8 using IBD-F fatigue score | 8 weeks
  Scored using a series of 35 questions, each scored from 0 to 4. The higher the total score (out of a possible total of 140), the higher the severity of fatigue.
Assessment of possible drug-related side effects: nausea, diarrhoea, mood disturbance, sleep disturbance - will all be assessed at baseline and week 8. | 8 weeks
  Measured using a binary outcome (yes/no) measure when asked whether any of the aforementioned symptoms have been experienced by the participant during the study period.

OTHER OUTCOMES:
Experimental arm 1: Assessment of faecal metabolome composition at baseline and week 8 | 8 weeks
  Faecal metabolome will be assessed by analysing the faecal headspace volatile organic compounds using semi-quantitative solid-phase microextraction gas chromatography mass spectrometry. Data will be presented using the relative abundance metrics for the key metabolites identified.
Experimental arm 2: Assessment of faecal microbiota composition at baseline and week 8 | 8 weeks
  Faecal microbiome will be assessed using high throughput metagenomic sequencing. Data will be presented using relative abundance metrics for the key microbes identified.

CONTACTS AND LOCATIONS:
Overall Officials: T Conley, Principal Investigator — Liverpool University Foundation NHS Trust
Locations (1):
- Liverpool University Foundation NHS Trust, Liverpool, United Kingdom

REFERENCES:
- [Background] Kulnigg S, Gasche C. Systematic review: managing anaemia in Crohn's disease. Aliment Pharmacol Ther. 2006 Dec;24(11-12):1507-23. doi: 10.1111/j.1365-2036.2006.03146.x. PMID 17206940
- [Background] Gasche C, Berstad A, Befrits R, Beglinger C, Dignass A, Erichsen K, Gomollon F, Hjortswang H, Koutroubakis I, Kulnigg S, Oldenburg B, Rampton D, Schroeder O, Stein J, Travis S, Van Assche G. Guidelines on the diagnosis and management of iron deficiency and anemia in inflammatory bowel diseases. Inflamm Bowel Dis. 2007 Dec;13(12):1545-53. doi: 10.1002/ibd.20285. PMID 17985376
- [Background] Hodges P, Gee M, Grace M, Thomson AB. Vitamin and iron intake in patients with Crohn's disease. J Am Diet Assoc. 1984 Jan;84(1):52-8. PMID 6690565
- [Background] Gisbert JP, Gomollon F. Common misconceptions in the diagnosis and management of anemia in inflammatory bowel disease. Am J Gastroenterol. 2008 May;103(5):1299-307. doi: 10.1111/j.1572-0241.2008.01846.x. PMID 18477354
- [Background] Stein J, Hartmann F, Dignass AU. Diagnosis and management of iron deficiency anemia in patients with IBD. Nat Rev Gastroenterol Hepatol. 2010 Nov;7(11):599-610. doi: 10.1038/nrgastro.2010.151. Epub 2010 Oct 5. PMID 20924367
- [Background] Schroder O, Mickisch O, Seidler U, de Weerth A, Dignass AU, Herfarth H, Reinshagen M, Schreiber S, Junge U, Schrott M, Stein J. Intravenous iron sucrose versus oral iron supplementation for the treatment of iron deficiency anemia in patients with inflammatory bowel disease--a randomized, controlled, open-label, multicenter study. Am J Gastroenterol. 2005 Nov;100(11):2503-9. doi: 10.1111/j.1572-0241.2005.00250.x. PMID 16279906
- [Background] Erichsen K, Ulvik RJ, Nysaeter G, Johansen J, Ostborg J, Berstad A, Berge RK, Hausken T. Oral ferrous fumarate or intravenous iron sucrose for patients with inflammatory bowel disease. Scand J Gastroenterol. 2005 Sep;40(9):1058-65. doi: 10.1080/00365520510023198. PMID 16165718
- [Background] Kulnigg S, Stoinov S, Simanenkov V, Dudar LV, Karnafel W, Garcia LC, Sambuelli AM, D'Haens G, Gasche C. A novel intravenous iron formulation for treatment of anemia in inflammatory bowel disease: the ferric carboxymaltose (FERINJECT) randomized controlled trial. Am J Gastroenterol. 2008 May;103(5):1182-92. doi: 10.1111/j.1572-0241.2007.01744.x. Epub 2008 Mar 26. PMID 18371137
- [Background] Lindgren S, Wikman O, Befrits R, Blom H, Eriksson A, Granno C, Ung KA, Hjortswang H, Lindgren A, Unge P. Intravenous iron sucrose is superior to oral iron sulphate for correcting anaemia and restoring iron stores in IBD patients: A randomized, controlled, evaluator-blind, multicentre study. Scand J Gastroenterol. 2009;44(7):838-45. doi: 10.1080/00365520902839667. PMID 19330567
- [Background] Munoz M, Villar I, Garcia-Erce JA. An update on iron physiology. World J Gastroenterol. 2009 Oct 7;15(37):4617-26. doi: 10.3748/wjg.15.4617. PMID 19787824
- [Background] Hallberg L, Ryttinger L, Solvell L. Side-effects of oral iron therapy. A double-blind study of different iron compounds in tablet form. Acta Med Scand Suppl. 1966;459:3-10. doi: 10.1111/j.0954-6820.1966.tb19403.x. No abstract available. PMID 5957969